CLINICAL TRIAL: NCT03129373
Title: Clinical Trial to Demonstrate the Comparative Efficacy of a Cryogenic Treatment (Medical Device) In Common and Plantar Warts Management
Brief Title: Clinical Study : Efficacy and Safety of Three Cryotherapy Devices for Wart Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oystershell NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14E2344
Record Dates: First submitted 2017-04-03; First posted 2017-04-26 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Warts
MeSH Terms: conditions — Warts

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pixie group (Experimental): Cryogenic treatment of wart (liquified nitrous oxide)
  * Maximum 3 application by the technician in charge of the study.
  * Apply between 15 to 20 sec on hand and 40 sec on feet.
  Interventions: Device: Cryogenic treatment of warts
- Wartner group (Active Comparator): Cryogenic treatment of wart (dimethylether propane-based):
  * Maximum 3 application by the technician in charge of the study.
  * Apply between 15 to 20 sec on hand and 40 sec on feet.
  Interventions: Device: Cryogenic treatment of warts
- Wortie group (Active Comparator): Cryogenic treatment of wart (dimethylether-based product):
  * Maximum 3 application by the technician in charge of the study.
  * Apply between 15 to 20 sec on hand and 40 sec on feet.
  Interventions: Device: Cryogenic treatment of warts

INTERVENTIONS:
Device: Cryogenic treatment of warts — Treatment of common and plantar wart by cryotherapy treatment.

SUMMARY:
The present study was set-up to evaluate clinical efficacy of Pixie® cryogenic pen versus two comparator cryogenic products (Wartner® and Wortie®) for the treatment of common and plantar warts.

DETAILED DESCRIPTION:
The use of cryotherapy has been long known to be effective against warts. The indications for Pixie® are in line with the indications presented in the collected literature data, as well as with the indications of equivalent devices.

The benefits of warts treatment without the use of chemicals are clearly evidenced. The treatment period is much shorter (one treatment compared to daily application of keratinolytics or fluorouracil, over a period of a few weeks). The cryogen therapy application through a conic tip is much more precise than with chemical substances. Chemical substance application is leading to more side effects of the surrounding skin (typical for chemical treatment are pain, blistering, ulceration and contact dermatitis).

The Instructions for Use were developed in line with these data and are therefore covering all hazards known up to the date of this report.

Based on these data the product received its CE-mark approval

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject.
* Sex: male or female.
* Age: more than 4 years old.
* Subject presenting at least 1 new common wart on hand or on feet or plantar wart (wart present since less than 6 months).
* Subject, including minors aged more than 14 years, having given freely and expressly his/her informed consent.
* Minor whose legal guardians have given their free and express informed consent.
* Subject who is able to comply with the study requirements, as defined in the present protocol, at the Investigator's appreciation.
* Subject able to comply with protocol requirements, as defined in the protocol.
* Subject or child's legal guardians being affiliated to a health social security system.
* Female subjects of childbearing potential should use a medically accepted contraceptive regimen (at the Investigator's discretion) since at least 12 weeks before the beginning of the study, during all the study.

Exclusion Criteria:

* Pregnant, parturient or nursing woman or planning a pregnancy during the study.
* Subject who had been deprived of their freedom by administrative or legal decision.
* Subject in a social or sanitary establishment.
* Major subject who is under guardianship or who is not able to express his consent.
* Subject suspected to be non-compliant according to the Investigator's judgment.
* Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results.
* Subject with a cutaneous disease other than common and plantar warts, on the studied zone.
* Subject with a known allergy to one of the component of the products or to the comparator.
* Subject who has diabetes.
* Subject having problems with blood circulation, or having a blood clotting condition.
* Subject with immune deficiency or autoimmune disease.
* Subject presenting more than 10 warts on the body.
* Subject presenting bleeding warts.
* Subject presenting birthmarks, moles, warts with hairs growing from them, or any other spots.
* Subject having a sensitive skin, inflamed, infected, irritated, red, damaged, cut, grazed, diseased or itchy on the treated zone.
* Subject presenting genital warts, flat warts, filiform warts, periungual warts or warts larger than 0.8cm.
* Subject undergoing a topical treatment on the test area or a systemic treatment:
* immunosuppressors and/or corticoids during the 4 previous weeks and during the study,
* retinoids during the 6 previous months and during the study,
* any medication stabilized for less than one month.
* Subject who received a treatment of any type on the selected wart during the previous 6 months.
* Intensive exposure to sunlight or UV-rays on the studied zone within the previous month and/or foreseen during the study.
* Subject planning to change her/his life habits during the study.
* Subjects must not take part in any other clinical study whilst taking part in this study.
* Subjects must not deliberately "sunbathe" for the duration of the study on the studied zone in case they cannot cover the treated area from sunlight.
* No product (except usual hygiene products and except for the prescribed after treatment) is to be used on the selected wart during the study. The subjects will continue to use their usual hygiene products, but they must not change the brand or use new products throughout the course of the study.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Comparison of the percentage of subjects with clinical wart remission after 1 treatment in the Pixie® group versus comparators groups (Wartner® and Wortie®), as observed during a clinical evaluation of the treated wart by the dermatologist. | After 1 treatment (approximately 15 days after the first treatment)

SECONDARY OUTCOMES:
Comparison of the number of treatments needed for clinical remission of warts with the three products. | 1 treatment (day 0), 2 treatments (day 15), 3 treatments (day 29)
Surface area measurements of frostbite area to evaluate the efficacy of the freezing process, during the three applications if applicable. | 1 treatment (day 0), 2 treatments (day 15), 3 treatments (day 29)
  Measurement immediately after treatment, with a tape measure device of the frostbite on the skin, created by cryothereapy treatment (measure in cm)
Illustration of the visual aspects of the wart remission with macrophotographs. | Before treatment (day 0 before treatment), after 1 treatment (day 15), after 2 treatments (day 29), after 3 treatments (day 45)
  Macrophotographs taken with a Nikon D90 apparatus and a standardization device for the repositionning
Evaluation of the skin conditions at study end, assessed by the investigator by clinical evaluation. | Before treatment (day 0 before treatment), after 1 treatment (day 15), after 2 treatments (day 29), after 3 treatments (day 45)
  Evaluation of the skin color after treatment.
Recording of adverse events. | On days 0, 3, 15, 29 and 45
Comparison of the percentage of subjects with clinical wart remission after 1, 2 and 3 treatments in the Pixie® group versus comparators groups (Wartner® and Wortie®), as observed during a clinical evaluation of the treated wart by the dermatologist. | After 1 treatment (day 15), after 2 treatments (day 29), after 3 treatments (day 45)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walczuk I, Eertmans F, Rossel B, Cegielska A, Stockfleth E, Antunes A, Adriaens E. Efficacy and Safety of Three Cryotherapy Devices for Wart Treatment: A Randomized, Controlled, Investigator-Blinded, Comparative Study. Dermatol Ther (Heidelb). 2018 Jun;8(2):203-216. doi: 10.1007/s13555-017-0210-5. Epub 2017 Dec 6. PMID 29214505